CLINICAL TRIAL: NCT05503563
Title: A Proposed Tetra-modal Treatment Protocol for Muscle Invasive Urothelial Carcinoma of the Urinary Bladder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Atef Ali, Urologist at Assuit University Hospital, Assiut University
Other Study IDs: AssuitUUro
Record Dates: First submitted 2022-07-29; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Bladder Cancer
Keywords: Tetramodal bladder preservation; urothelial carcinoma; partial cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- tetra modal bladder preservation
  Interventions: Procedure: terta modal bladder preservation

INTERVENTIONS:
Procedure: terta modal bladder preservation — neoadjuvant chemotherapy, partial cystectomy, radiotherapy

SUMMARY:
In Egypt, bladder cancer has been the most common cancer during the past 50 years. In 2002, Egypt's world-standardized bladder cancer incidence was 37/ 100,000, representing approximately 30,000 new cases each year.

About 25% of new diagnoses are muscle-invasive bladder cancer (MIBC), which carry a worse prognosis compared to non-muscle invasive disease.

Neoadjuvant chemotherapy (NAC) followed by radical cystectomy (RC) with bilateral pelvic lymphadenectomy is considered the standard of care for treatment of MIBC by multiple international guidelines.

However, this is associated with a significant impact on quality of life.

The effect of our proposed Tetra-modal treatment protocol for muscle invasive Urothelial carcinoma of the urinary bladder on muscle invasive bladder cancer recurrence free survival, cancer specific survival, and overall survival?

Koga developed a selective bladder-sparing protocol with a tetra modal therapy comprising maximal transurethral resection of bladder tumor, induction chemoradiation (CRT), and consolidative partial cystectomy (PC) with pelvic lymph node dissection, allowing the confirmation of CRT response pathologically. In the preliminary analysis of the initial cases enrolled in their protocol, none of the patients who completed the protocol with consolidative PC experienced MIBC recurrence, suggesting that consolidative PC may improve local cancer control in the preserved bladder by surgically eliminating possible cancer remnants after CRT.

Our proposed Tetra-modal treatment protocol for MIBC is supposed to eliminate the surgical difficulties of performing PC in a radiated field and hence decrease the post operative complications of PC.

ELIGIBILITY:
Inclusion Criteria:

1. Tumor size ≤ 50 % of bladder surface or multiple tumors in an area of the bladder that is ≤ 50 % of total bladder surface.
2. Tumor at least 2 cm away from bladder neck or trigone.
3. Clinically, no residual disease or minimal amounts of non-invasive disease in the original MIBC site after NAC at restaging TURBT (if done).
4. Pathologically confirmed urothelial carcinoma.

Exclusion Criteria:

1. Prescence of CIS.
2. Presence of distant metastasis.
3. Patients unfit for cisplatin-based chemotherapy.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient presented with bladder cancer whom are under treatment with multiple modalities such as endoscopic resection , chemotherapy , radiotherapy & partial cystectomy,
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
local recurrence rate | the patient will be evaluted after partial cystectomy every 3 months for 2 years
  the patient will be evaluated using MRI and cystoscopy
over active bladder symptom score | this questionnaire will be carried every 6 month for at least 2 years after the partial cystectomy
  the patient will be asked about his symptoms using a questionnaire that is concerned about urgency , frequency , urge incontinence .

CONTACTS AND LOCATIONS:
Overall Officials: Diaa A Sayed, PhD, Study Director — cheif of urological oncology department
Locations (1):
- Assuit university, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Felix AS, Soliman AS, Khaled H, Zaghloul MS, Banerjee M, El-Baradie M, El-Kalawy M, Abd-Elsayed AA, Ismail K, Hablas A, Seifeldin IA, Ramadan M, Wilson ML. The changing patterns of bladder cancer in Egypt over the past 26 years. Cancer Causes Control. 2008 May;19(4):421-9. doi: 10.1007/s10552-007-9104-7. Epub 2008 Jan 10. PMID 18188671
- [Background] Burger M, Catto JW, Dalbagni G, Grossman HB, Herr H, Karakiewicz P, Kassouf W, Kiemeney LA, La Vecchia C, Shariat S, Lotan Y. Epidemiology and risk factors of urothelial bladder cancer. Eur Urol. 2013 Feb;63(2):234-41. doi: 10.1016/j.eururo.2012.07.033. Epub 2012 Jul 25. PMID 22877502
- [Background] Kulkarni GS, Black PC, Sridhar SS, Kapoor A, Zlotta AR, Shayegan B, Rendon RA, Chung P, van der Kwast T, Alimohamed N, Fradet Y, Kassouf W. Canadian Urological Association guideline: Muscle-invasive bladder cancer. Can Urol Assoc J. 2019 Aug;13(8):230-238. doi: 10.5489/cuaj.5902. No abstract available. PMID 30763236
- [Background] Noone AM, Cronin KA, Altekruse SF, Howlader N, Lewis DR, Petkov VI, Penberthy L. Cancer Incidence and Survival Trends by Subtype Using Data from the Surveillance Epidemiology and End Results Program, 1992-2013. Cancer Epidemiol Biomarkers Prev. 2017 Apr;26(4):632-641. doi: 10.1158/1055-9965.EPI-16-0520. Epub 2016 Dec 12. PMID 27956436
- [Background] Singh AK, Shukla PK, Khan SW, Rathee VS, Dwivedi US, Trivedi S. Using the Modified Clavien Grading System to Classify Complications of Percutaneous Nephrolithotomy. Curr Urol. 2018 Feb;11(2):79-84. doi: 10.1159/000447198. Epub 2017 Dec 30. PMID 29593466